CLINICAL TRIAL: NCT00157586
Title: A Multicenter, Randomized, Prospective, Double-blind Study to Evaluate the Nephroprotective Effect of Delapril Alone or Combined With Manidipine in Patients With Type 2 Diabetes
Brief Title: Delapril and Manidipine for Nephroprotection in Diabetes (DEMAND)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DM/PR/7401/005/00
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2006-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — delapril

INTERVENTIONS:
Drug: Delapril, Delapril-Manidipine Fixed combination

SUMMARY:
Diabetes mellitus is one of the most common diseases globally, and is considered epidemic in many developed and newly industrialized nations. Diabetes mellitus represents the single largest cause of end-stage renal disease in the U.S. and Europe. At the same time, the primary cause of early death in diabetic patients are cardiovascular complications. Experimental and clinical studies found that angiotensin converting enzyme inhibitors (ACEi) and calcium channel blockers (CCBs) have a specific renoprotective effect and that this effect can be magnified when the two drugs are used in combination. To formally test this hypothesis we designed the Delapril and Manidipine for Nephroprotection in Diabetes (DEMAND) study, a prospective, randomized, double blind trial aimed to compare the effect of 3 years treatment with the ACEi Delapril (30 mg/day), alone or combined to the CCB Manidipine (10 mg/day), versus conventional (non ACEi, non CCB) therapy on the rate of renal function loss and on the incidence of major cardiovascular events in 342 normo- and micro-albuminuric hypertensive type 2 diabetic patients.

DETAILED DESCRIPTION:
INTRODUCTION Optimal blood pressure, glycemic and lipid control are of utmost importance to minimize the incidence and the progression of chronic renal and cardiovascular complications in patients with diabetes mellitus type 2. Whether angiotensin converting enzyme (ACE) inhibitors alone or combined to calcium channel blockers (CCB) may further reduce the incidence and progression of chronic complications is worth investigating.

AIMS The primary aim of this study is to assess whether at comparable levels of optimal blood pressure and metabolic control, the ACE inhibitor delapril alone or in combination with the dihydropyridine CCB manidipine slow the rate of glomerular filtration rate (GFR) decline as compared with placebo plus conventional antihypertensive therapy in patients with diabetes mellitus type 2 and hypertension. The secondary aim of this study is to assess the effects of delapril and manidipine on the incidence of major cardiovascular events (acute myocardial infarction, ictus or stroke, heart failure requiring hospitalization, revascularization, amputation and cardiovascular mortality).

STUDY POPULATION 342 hypertensive type 2 diabetes patients with normo- or micro-albuminuria. STUDY DESIGN This is a multicenter, prospective, randomized, double-blind, placebo-controlled study. After a 12-week baseline period in which prohibited antihypertensive treatments (ACE inhibitors, angiotensin II receptor antagonists or dihydropyridine calcium channel blockers) will be discontinued, patients will be stratified according to their urinary albumin excretion rate in normo- and micro-albuminuric and then randomized to delapril alone (30 mg/day), delapril (30 mg/day) combined with manidipine (10 mg/day) or placebo given once daily in the morning for at least three years. During the study, systolic and diastolic blood pressure in all treatments groups will be maintained ≤ 120 and 80 mmHg respectively, with fixed doses of study treatments and flexible doses of permitted antihypertensive therapy (diuretics, beta blockers, alfa blockers, centrally acting adrenergic blockers. Blood pressure, blood glucose concentrations and urinary albumin excretion rate will be monitored every three months. Serum lipid concentrations and GFR (estimated with the iohexol plasma clearance) will be measured every six months.

Primary and Secondary Variables. The primary efficacy variable of this study is the rate of GFR decline. The secondary efficacy variable will be the incidence of major cardiovascular events (acute myocardial infarction, ictus or stroke, heart failure requiring hospitalization, revascularization, amputation and cardiovascular mortality).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* History of diabetes mellitus type 2 for at least three months with stable antidiabetic treatment
* Systolic and/or diastolic blood pressure ≥ 135 or 85 mmHg, respectively. In alternative, antihypertensive therapy regardless of blood pressure values
* Serum creatinine ≤ 1.5 mg/dL
* Urinary albumin excretion rate < 200 µg/min
* Written informed consent for the trial participation.

Exclusion Criteria:

* Clinical or histological evidence of non-diabetic renal disease, including vascular disease of the kidney, obstructive uropathy, prostatic hypertrophy or incomplete bladder emptying
* Transplanted kidney
* Moderate to severe chronic heart failure (III-IV stage according to the NYHA classification).
* Cerebral hemorrhage, stroke or transient ischemic attack within three months prior to the trial enrolment
* Myocardial infarction within three months prior to the trial enrolment
* Unstable angina pectoris
* Mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
* Secondary (e.g., Cushing disease, phaeochromocytoma, etc.) or severe refractory hypertension
* Poor glycemic control (HbA1c>11%)
* Connective tissue or autoimmune disease
* Hereditary angioneurotic edema
* Clinically relevant electrolyte imbalance (e.g., serum potassium > 5.5 mmol/L)
* Clinically relevant hematological disorders
* Anemia with hemoglobin concentrations < 10 g/dL
* Serious hepatic disease
* Pregnancy or lactating or planning a pregnancy
* Women of childbearing potential without following a scientifically accepted form of contraception
* Any other serious or terminal concomitant disease
* Any condition which may interfere with the absorption of the study treatments
* Any concomitant treatment with ACE inhibitors, angiotensin II blockers, calcium channel blockers, potassium sparing diuretics
* Chronic treatment with nonsteroidal antiinflammatory drugs, antidepressants and neuroleptics, lithium, cimetidine, immunosuppressive and/or antineoplastic drugs, chronic systemic glucocorticoid therapy more than 7 consecutive days in one month, antiarrhythmic drugs (e.g., chinidin, procainamide), anesthetics/narcotics
* History of hypersensitivity to delapril or other ACE inhibitors, manidipine or other dihydropyridine CCBs
* Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequences of the trial
* Evidence of an uncooperative attitude
* Any evidence that allows predicting that the patient will not be able to complete the trial follow-up.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342
Dates: Start 2002-02; Study Completion 2008-06

PRIMARY OUTCOMES:
The rate of decline of glomerular filtration rate (GFR).GFR is measured at baseline,and at 6,12,18,24,30 and 36 months after randomization

SECONDARY OUTCOMES:
Major cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ruggenenti, MD, Principal Investigator — Mario Negri Institute
Locations (8):
- Italy (7):
  - Hospital "Ospedali Riuniti di Bergamo" - Diabetologic Unit, Bergamo, Bergamo
  - ASL of Ponte San Pietro - Diabetologic Unit, Ponte San Pietro, Bergamo
  - Clinical Research Center for Rare Diseases, Ranica, Bergamo
  - Hospital of Romano di Lombardia - Diabetologic Unit, Romano di Lombardia, Bergamo
  - Hospital " Bolognini " - Medicine Unit, Seriate, Bergamo
  - Hospital " Treviglio Caravaggio" - Diabetologic Unit, Treviglio, Bergamo
  - Humanitas Institute - Endocrinology and Diabetologic Unit, Rozzano, Milano
- Department of Endocrinolgy, Diabetes and Metabolic Disease - University Medical Center, Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Carrara F, Ruggenenti P, Perna A, Iliev IP, Gaspari F, Ferrari S, Stucchi N, Bossi A, Trevisan R, Remuzzi G, Parvanova A. Glomerular resistances predict long-term GFR decline in type 2 diabetic patients without overt nephropathy: a longitudinal subgroup analysis of the DEMAND trial. Acta Diabetol. 2022 Mar;59(3):309-317. doi: 10.1007/s00592-021-01804-9. Epub 2021 Oct 14. PMID 34648087
- [Derived] Ruggenenti P, Porrini EL, Gaspari F, Motterlini N, Cannata A, Carrara F, Cella C, Ferrari S, Stucchi N, Parvanova A, Iliev I, Dodesini AR, Trevisan R, Bossi A, Zaletel J, Remuzzi G; GFR Study Investigators. Glomerular hyperfiltration and renal disease progression in type 2 diabetes. Diabetes Care. 2012 Oct;35(10):2061-8. doi: 10.2337/dc11-2189. Epub 2012 Jul 6. PMID 22773704
- [Derived] Ruggenenti P, Lauria G, Iliev IP, Fassi A, Ilieva AP, Rota S, Chiurchiu C, Barlovic DP, Sghirlanzoni A, Lombardi R, Penza P, Cavaletti G, Piatti ML, Frigeni B, Filipponi M, Rubis N, Noris G, Motterlini N, Ene-Iordache B, Gaspari F, Perna A, Zaletel J, Bossi A, Dodesini AR, Trevisan R, Remuzzi G; DEMAND Study Investigators. Effects of manidipine and delapril in hypertensive patients with type 2 diabetes mellitus: the delapril and manidipine for nephroprotection in diabetes (DEMAND) randomized clinical trial. Hypertension. 2011 Nov;58(5):776-83. doi: 10.1161/HYPERTENSIONAHA.111.174474. Epub 2011 Sep 19. PMID 21931073